CLINICAL TRIAL: NCT03647254
Title: Effectivity of a Joint Didactic Intervention by School for Patients on Inappropriate Control Prothrombin Time Anticoagulated Patients. Protocol for Developing a Randomized and Controlled Clinical Trial
Brief Title: Efficacy of a Didactic Intervention in Anticoagulated Patients (TAOPE Study)
Acronym: TAOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Francisco Javier Navarro Moya (Other Government)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Sponsor-Investigator, Francisco Javier Navarro Moya, Effectiveness and Research Unit Coordinator. District of Malaga. Andalusian Health Service. Spain, Andaluz Health Service
Organization: Andaluz Health Service (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AndaluzHS
Record Dates: First submitted 2018-08-08; First posted 2018-08-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Health Education; Patient Education as Topic; Blood Coagulation Tests
Keywords: Anticoagulants; Warfarin
MeSH Terms: conditions — Health Education | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education Group (Experimental): A group educational intervention was practiced to half of the patients, by one expert patient, so that every patient must attend to one group meeting and they continued with their usual controls
  Interventions: Behavioral: Patient education group
- Control group (No Intervention): Control group performed usual clinical practice, that is, people will be schedule by nurses about one time per month, except cases in which controls are inappropriate.

INTERVENTIONS:
Behavioral: Patient education group — Group meetings with educational sessions will be organised in health center. A group educational intervention was practiced to half of the patients, by one expert patient, so that every patient must attend to one group meeting
  Other Names: Control group
  Arms: Patient Education Group

SUMMARY:
Background: Oral anticoagulant drugs represent an essential tool in thrombo-embolic events prevention. Most used are vitamin K antagonists (VKA), which plasma level is monitored measuring prothrombin time using the International Normalized Ratio. If it takes values out of recommended range, the patient will have a higher risk of suffering from thromboembolic or hemorrhagic complications. Previous researches have shown that, at best, only 33% of total patients keep values on therapeutic level.

The investigators intend to improve International Normalized Ratio control figures by a joint didactic intervention based on Junta de Andalucía School for Patients method that will be practiced by anticoagulated patients themselves.

Methods: A randomized clinical trial was carried out at primary care centers from one healthcare area in Malaga (Andalusia, Spain). Study population: patients included on oral anticoagulant therapy program using vitamin K antagonists.

First step: detection of patients on oral anticoagulation program with International Normalized Ratio on therapeutic level during 65% or less over total time. Second step: patients with inappropriate International Normalized Ratio control were practiced a joint didactic intervention "from peer to peer", by a previously trained and expert anticoagulated patient.

Study variables: time on therapeutic levels before and after intervention, sociodemographic variables, vital signs, existence of cardiovascular risk factors, basic blood test, other prescribed drugs, accompanying diseases and social support.

Almost-experimental analytic study with before-after statistical analysis of the intervention. Lineal regression models were applied on main variables results (International Normalized Ratio value, time on therapeutic level) inputting sociodemographic variables, accompanying diseases and social support.

DETAILED DESCRIPTION:
Background and current status:

It has been proved that oral anticoagulant therapy (OAT) is effective in preventing situations with high risk of thromboembolic events and in treating them. It significantly decreases ischemic stroke rates as well as their severity and death risk. However it is a therapy with special features, highlighting: doses and response variability, the close therapeutic range, interactions with other drugs and foods, and potentially severe side effects. This fact compels the investigators to make a close monitoring of those patients.

An important impact in developing cardioembolic or hemorrhagic events due to a inappropriate coagulation control using vitamin K antagonists (VKA), has been described; because of control variations around 15% could result in so relevant clinical problems.

The main OAT indications are deep vein thrombosis, pulmonary embolism, embolic conditions prevention in patients suffering from atrial fibrillation or heart prosthetic valve wearers. Most common embolic event is ictus, which could lead to an important inability and dependence state, what would associate a significant increase in health resources use and costs. Atrial fibrillation (AF) is nowadays the pathology which requires most anticoagulant therapy indications. This fact is partially due to the population aging, since there are both incidence and prevalence increases of this arrhythmia, specially in elderly patients.

Control of patients on OAT were performed in hospitals until a few years ago; nevertheless, changes in social and healthy contexts besides the expansion in this drugs prescribing joined to primary health care qualification and evolution, the development of coagulation handheld measuring devices and the need to improve patients accessibility, had justified the control decentralization and due to this facts, OAT monitoring can be practiced to stable patients on primary care.

When the need of receiving anticoagulation has been stablished, this could be implemented basically using heparin or vitamin-K antagonists or coumadin or new direct action oral anticoagulants as dabigatran, rivaroxaban, apixaban or edoxaban.

The prothrombin time measuring standardization using international normalized ratio (INR) allows the investigators to obtain reliable results in different laboratories. The development of coagulation handheld measuring devices to match INR in capillary blood with high sensitivity and reliability, has made that possible patients on anticoagulant therapy can be controlled on primary care. This allow the investigators a comprehensive approach and control of these patients.

Educational and behavioural interventions could improve VKA anticoagulated patients ability to keep an INR appropriate control using their progresses in knowledge and understanding of the action mechanisms of anticoagulants drugs. A recent research included in Cochrane regarding to those interventions notes that education is particularly important to provide information about safety for patients suffering AF on OAT and let patients to take their own well founded decisions about treatment options and to manage their OAT. However, it could be inferred there are not enough evidences to stablish definite conclusions about educational health interventions impact in INR behaviour in patients suffering from AF on OAT.

In the investigators environment, patients who initiate treatment with VKA are trained at their hematology units until they get a suitable INR level control. After that, patients are followed and evaluated in primary care. The amount of patients with AF on anticoagulation with VKA is high, however, INR levels control results are not ideal.

Therefore, in these three research articles recently conducted in Spain with patients on VKA, it can be observed an inappropriate anticoagulation control.

On the other hand, it should be noted that these chronic patients use to suffer many other conditions and they usually take a lot of medication which makes improve of education aspects aimed at self care and effective health self-management which is absolutely necessary. Selfcare support programs are presented as a tool to accomplish a change in paternalistic method to other one in which citizens could receive more information about their health state (this fact is in accordance with people requests, demonstrated by a rise in the internet consulting about health issues).

"Expert patients" programs, in which instructors are patients with chronic conditions similar to those who receive the training and so they could play a role model, occupying a prominent place inside the selfcare educational initiatives set.

Through the present research the investigators try to show that an organised group educational intervention, conducted by using School for Patients method on VKA anticoagulated patients is able to improve inappropriate INR levels control.

METHODS:

The investigators performed a randomized clinical trial over a period of 12 months.

Study area: one healthcare area in Malaga (Spain) where 741.000 inhabitants from rural or urban population are cared for. It is organized in 33 primary care centers and 19 local doctor´s offices.

Study population: patients on OAT program receiving VKA presenting inappropriate INR levels control and belonging to four primary care centers. Setting the limits and justification of the sample size:

Total population from the health centers which take part in the study amount to approximately 50.000 inhabitants.

Step I: If it is taken into account that prevalence of patients on OAT is about 1.5% of general population, it can be claimed that target population to initiate the study will be 750 anticoagulated patients. It has been observed in previous researches that at least 33% of these patients would not have an appropriate INR level control. In order to reach an accuracy about 4% in the estimate proportion using a normal asymptotic confidence interval with a correction to finite populations on bilaterally 95% and assuming that expected population is about 33% and population total size is 750, it will be necessary to include 311 experimental units in this study.

Step II: If it is accepted an alfa risk of 0.05 and a beta risk of 0.20 in a bilateral contrast between study group and control group, 312 individual will be required (156 in each group) to detect differences equal or higher than 15% between both groups in primary target. It has been estimated a tracking loss rates of 10%. It will be assumed as losts those individual impossible to be located, or those who do not accept to take part or those who do not attend to scheduled revisions, in accordance to the study intervention plan, as well as deceases occurring within six months since the intervention. Given the relevant impact of the development of cardioembolic or hemorrhagic events due to inappropriate INR control, changes about 15% could have great clinical relevance.

Variables. Operative definition The main variable to assess in this study is time on INR therapeutic levels in the last six months receiving VKA treatment. Appropriate INR level control will be assessed in two ways: measuring the therapeutic INR values percentages or Time percentages in therapeutic values estimated using Rosendaal method. It supposes to record the figure of INR value and the date in which the test was carried out. The therapeutic INR values percentages are defined by their acceptable values according to the pathology the patient suffers. It used to be from 2 to 3 if it is about atrial fibrillation or from 2.5 to 3.5 if thromboembolism prevention is carried out after a heart valve surgery has been performed. So, this quantitative variable has to be measured to calculate patients percentage on appropriate range, according to the patient condition.

Independent variables also called study variables are those which could affect to result variable. The investigators are going to classify them in eight groups to make easier their analysis.

Sociodemographic: age and gender. Somatometry and vital signs: Body mass index (BMI), diastolic and systolic blood pressure, and heart rate.

Cardiovascular risk factors: smoking habit, diabetes, arterial hypertension, dyslipidemia and chronic renal failure.

Cardiovascular conditions: atrial fibrillation (AF), interventional cardiac valve diseases with or without AF, ischemic cardiopathy, thromboembolic diseases history (stroke, transient ischemic attack), hemorrhagic stroke, congestive heart failure.

Blood test: Glomerular filtration rates, total cholesterol, HDL and LDL cholesterol and triglycerides. They will be obtained from the last blood test carried out to the patient.

Use of accompanying medication: total number of drugs, anticoagulant type. Consumption of "gastric protector".

Dietary habits: usual consumption of food rich in vitamin K, alcohol consumption.

Data collecting: All variables detailed previously were collected as long as they were suitable in digital medical history or it could be directly obtained from the patient during the medical interview, without the need of changing health center usual clinical practice, over the 6 months prior to the intervention.

First step: patients on OAT program enrolled in several primary health centers belonging to a healthcare area of Málaga were evaluated at the study moment attending to their clinical characteristics. The measurements obtained from the digital clinical history in the last six months before the beginning of the study were recorded, as well as the rest of variables.

Second step: Once the study of the VKA anticoagulation control degree has been performed, patients on inappropriate control were selected. A list of patients with deficient INR control in participant health centers was made. It was considered an inappropriate INR control when the therapeutic INR values percentages was less than 65%, using Rosendaal method to obtain them. In case of no availability, INR control was considered inappropriate when therapeutic INR values percentage resulted less than 60%. In any of the assumptions, the assessment period was at least the last six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients on VKA treatment for at least the last six months in primary care environment.
* Patients on inappropriate INR level control.
* Patients in whom we have access to, at least, 80% of their INR levels. controls in last six months of treatment with VKA, although they are enrolled in another primary care center.
* Patients who have given written informed consent to take part in the study

Exclusion Criteria:

* Patients suffering from cognitive impairment wich prevents understanding what was written in the information sheet and informed consent.
* Limited mobility patients, terminal patients, alcoholism or drug addiction, severe psychiatric illness or any other reason which makes patients to be present at center´s meetings imposible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Time on INR therapeutic levels in the last six months receiving VKA treatment | Six months
  Appropriate INR level control will be assessed in two ways: measuring the therapeutic INR values percentages or Time percentages in therapeutic values estimated using Rosendaal method

SECONDARY OUTCOMES:
Sociodemographic | Six months
  Record of age and sex.
Body mass index (BMI) | 0 and 12 months.
  Determination of the body mass index calculated as the weight measured in kilograms (kg) divided by the height measured in meters squared (weight / height2) (Kg /m2).
Diastolic and systolic blood pressure | 0 and 12 months.
  Determination of diastolic and systolic blood pressure measured in millimeters of mercury (mm / Hg), average of 2 determinations.
Heart rate | 0 and 12 months.
  Determination of the number of heart beats per minute, average of 2 Determination of
Smoking habit | 0 and 12 months.
  Incidence of smoker's habit status in the electronic medical record.
diabetes | 0 and 12 months.
  Incidence of the condition of diabetes in the electronic medical record.
Arterial hypertension | 0 and 12 months.
  Incidence of diagnosis of hypertension in the electronic medical record.
Dyslipidemia | 0 and 12 months.
  Incidence of the diagnosis of dyslipidemia in the electronic medical record.
Chronic renal failure | 0 and 12 months.
  Incidence of the diagnosis of chronic renal failure in the electronic medical record.
Atrial fibrillation | 0 and 12 months.
  Incidence of diagnosis of atrial fibrillation in the electronic medical records of patients.
Interventional cardiac valve diseases with or without atrial fibrillation | 0 and 12 months.
  Incidence of diagnosis of interventional cardiac valve diseases in the electronic medical records of patients.
Ischemic cardiopathy | 0 and 12 months.
  Incidence of diagnosis of Ischemic cardiopathy in the electronic medical records of patients.
Thromboembolic diseases history (stroke, transient ischemic attack) | 0 and 12 months.
  Incidence of diagnosis of thromboembolic diseases history (stroke, transient ischemic attack) in the electronic medical records of patients.
Hemorrhagic stroke | 0 and 12 months.
  Incidence of diagnosis of hemorrhagic stroke in the electronic medical records of patients.
Congestive heart failure | 0 and 12 months.
  Incidence of diagnosis of congestive heart failure in the electronic medical records of patients.
Glomerular filtration rates | 0 and 12 months.
  Determination of total Glomerular filtration rates in mL/min/1,73 m2. Change of basal to 12 months.
Total cholesterol | 0 and 12 months.
  Determination of total cholesterol measured in milligrams per deciliter (mg/dl). Change of basal to 12 months.
HDL Cholesterol | 0 and 12 months.
  Determination of HDLc (high-density lipoprotein colesterol). LDLc measured in milligrams per deciliter (mg/dl)., (low-density lipoprotein colesterol). HDLc measured in milligrams per deciliter (mg/dl). Change of basal to 12 months.
LDL cholesterol | 0 and 12 months.
  Determination of LDLc (low-density lipoprotein colesterol). LDLc measured in milligrams per deciliter (mg/dl). Change of basal to 12 months.
Triglycerides | 0 and 12 months.
  Determination of total triglycerides measured in milligrams per deciliter (mg/dl). Change of basal to 12 months.
Total number of drugs | 0 and 12 months.
  Determination of the total number of different medications prescribed in the electronic medical records of patients. Change of basal to 12 months
Anticoagulant type | 0 and 12 months.
  Determination of the anticoagulant type prescribed in the electronic medical records of patients. Change at baseline and at 12 months.
Consumption of "gastric protector" | 0 and 12 months.
  Determination of the Consumption of "gastric protector" prescribed in the electronic medical records of patients. Change at baseline and at 12 months.
Usual consumption of food rich in vitamin K | 0 and 12 months.
  Change in usual consumption of food rich in vitamin K. Change at baseline and at 12 months
Alcohol consumption | 0 and 12 months.
  Change in usual Alcohol consumption. Change at baseline and at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Navarro Moya, Enfermera, Study Chair — Servicio de salud pública de Andalucía. Málaga, España
Locations (1):
- Distrito Sanitario Málaga. Servicio Andaluz de Salud, Málaga, Spain

REFERENCES:
- [Background] Ageno W, Gallus AS, Wittkowsky A, Crowther M, Hylek EM, Palareti G. Oral anticoagulant therapy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e44S-e88S. doi: 10.1378/chest.11-2292. PMID 22315269
- [Background] Oden A, Fahlen M, Hart RG. Optimal INR for prevention of stroke and death in atrial fibrillation: a critical appraisal. Thromb Res. 2006;117(5):493-9. doi: 10.1016/j.thromres.2004.11.025. Epub 2004 Dec 25. PMID 16517250
- [Background] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Background] Wan Y, Heneghan C, Perera R, Roberts N, Hollowell J, Glasziou P, Bankhead C, Xu Y. Anticoagulation control and prediction of adverse events in patients with atrial fibrillation: a systematic review. Circ Cardiovasc Qual Outcomes. 2008 Nov;1(2):84-91. doi: 10.1161/CIRCOUTCOMES.108.796185. Epub 2008 Nov 5. PMID 20031794
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren M, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; European Association for Cardiovascular Prevention & Rehabilitation (EACPR); ESC Committee for Practice Guidelines (CPG). European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Eur Heart J. 2012 Jul;33(13):1635-701. doi: 10.1093/eurheartj/ehs092. Epub 2012 May 3. No abstract available. PMID 22555213
- [Background] Wolowacz SE, Samuel M, Brennan VK, Jasso-Mosqueda JG, Van Gelder IC. The cost of illness of atrial fibrillation: a systematic review of the recent literature. Europace. 2011 Oct;13(10):1375-85. doi: 10.1093/europace/eur194. Epub 2011 Jul 14. PMID 21757483
- [Background] Gomez-Doblas JJ, Muniz J, Martin JJ, Rodriguez-Roca G, Lobos JM, Awamleh P, Permanyer-Miralda G, Chorro FJ, Anguita M, Roig E; OFRECE study collaborators. Prevalence of atrial fibrillation in Spain. OFRECE study results. Rev Esp Cardiol (Engl Ed). 2014 Apr;67(4):259-69. doi: 10.1016/j.rec.2013.07.014. Epub 2013 Nov 25. PMID 24774588
- [Background] Naccarelli GV, Varker H, Lin J, Schulman KL. Increasing prevalence of atrial fibrillation and flutter in the United States. Am J Cardiol. 2009 Dec 1;104(11):1534-9. doi: 10.1016/j.amjcard.2009.07.022. PMID 19932788
- [Background] Robert-Ebadi H, Le Gal G, Righini M. Use of anticoagulants in elderly patients: practical recommendations. Clin Interv Aging. 2009;4:165-77. doi: 10.2147/cia.s4308. Epub 2009 May 14. PMID 19503778
- [Background] Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest. 2010 Feb;137(2):263-72. doi: 10.1378/chest.09-1584. Epub 2009 Sep 17. PMID 19762550
- [Background] Olesen JB, Lip GY, Hansen ML, Hansen PR, Tolstrup JS, Lindhardsen J, Selmer C, Ahlehoff O, Olsen AM, Gislason GH, Torp-Pedersen C. Validation of risk stratification schemes for predicting stroke and thromboembolism in patients with atrial fibrillation: nationwide cohort study. BMJ. 2011 Jan 31;342:d124. doi: 10.1136/bmj.d124. PMID 21282258
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Steinberg BA, Piccini JP. Anticoagulation in atrial fibrillation. BMJ. 2014 Apr 14;348:g2116. doi: 10.1136/bmj.g2116. PMID 24733535
- [Background] Riley RS, Rowe D, Fisher LM. Clinical utilization of the international normalized ratio (INR). J Clin Lab Anal. 2000;14(3):101-14. doi: 10.1002/(sici)1098-2825(2000)14:33.0.co;2-a. PMID 10797608
- [Background] Cardenas Valladolid J, Mena Mateo J, Canada Dorado MM, Rodriguez Morales D, Sanchez Perruca L. [Implementation and improvement in a care program for the elderly on multiple medications in a primary care area]. Rev Calid Asist. 2009 Feb;24(1):24-31. doi: 10.1016/S1134-282X(09)70072-7. Epub 2009 Feb 23. Spanish. PMID 19369139
- [Background] Clarkesmith DE, Pattison HM, Lane DA. Educational and behavioural interventions for anticoagulant therapy in patients with atrial fibrillation. Cochrane Database Syst Rev. 2013 Jun 4;(6):CD008600. doi: 10.1002/14651858.CD008600.pub2. PMID 23736948
- [Background] Lobos-Bejarano JM, del Castillo-Rodriguez JC, Mena-Gonzalez A, Aleman-Sanchez JJ, Cabrera de Leon A, Baron-Esquivias G, Pastor-Fuentes A; en nombre de los Investigadores del Estudio FIATE (Situacion actual de la FIbrilacion auricular en ATencion primaria en Espana). [Patients' characteristics and clinical management of atrial fibrillation in primary healthcare in Spain: FIATE Study]. Med Clin (Barc). 2013 Oct 5;141(7):279-86. doi: 10.1016/j.medcli.2012.12.023. Epub 2013 May 15. Spanish. PMID 23683967
- [Background] Gallagher AM, Setakis E, Plumb JM, Clemens A, van Staa TP. Risks of stroke and mortality associated with suboptimal anticoagulation in atrial fibrillation patients. Thromb Haemost. 2011 Nov;106(5):968-77. doi: 10.1160/TH11-05-0353. Epub 2011 Sep 8. PMID 21901239
- [Background] Han SY, Palmeri ST, Broderick SH, Hasselblad V, Rendall D, Stevens S, Tenaglia A, Velazquez E, Whellan D, Wagner G, Heitner JF. Quality of anticoagulation with warfarin in patients with nonvalvular atrial fibrillation in the community setting. J Electrocardiol. 2013 Jan-Feb;46(1):45-50. doi: 10.1016/j.jelectrocard.2012.08.011. Epub 2012 Oct 11. PMID 23063241
- [Background] Barrios V, Escobar C, Prieto L, Osorio G, Polo J, Lobos JM, Vargas D, Garcia N. Anticoagulation Control in Patients With Nonvalvular Atrial Fibrillation Attended at Primary Care Centers in Spain: The PAULA Study. Rev Esp Cardiol (Engl Ed). 2015 Sep;68(9):769-76. doi: 10.1016/j.rec.2015.04.017. Epub 2015 Jul 11. PMID 26169326
- [Background] Cinza Sanjurjo S, Rey Aldana D, Gestal Pereira E, Calvo Gomez C; ANFAGAL (ANticoagulacion en pacientes con Fibrilacion Auricular en ambito de atencion primaria de GALicia) study. Degree of Anticoagulation Control in Patients With Atrial Fibrillation in Spain: Need to Minimize Biases and Contextualize Results. Response by Cinza Sanjurjo et al. Rev Esp Cardiol (Engl Ed). 2016 Mar;69(3):357-8. doi: 10.1016/j.rec.2015.12.005. Epub 2016 Jan 30. No abstract available. PMID 26839056
- [Background] Rosendaal FR, Cannegieter SC, van der Meer FJ, Briet E. A method to determine the optimal intensity of oral anticoagulant therapy. Thromb Haemost. 1993 Mar 1;69(3):236-9. PMID 8470047
- [Background] Anguita Sanchez M, Bertomeu Martinez V, Cequier Fillat A; CALIFA study researchers. Quality of Vitamin K Antagonist Anticoagulation in Spain: Prevalence of Poor Control and Associated Factors. Rev Esp Cardiol (Engl Ed). 2015 Sep;68(9):761-8. doi: 10.1016/j.rec.2014.11.019. Epub 2015 Mar 23. PMID 25814183
- [Background] Richards T, Montori VM, Godlee F, Lapsley P, Paul D. Let the patient revolution begin. BMJ. 2013 May 14;346:f2614. doi: 10.1136/bmj.f2614. No abstract available. PMID 23674136
- [Background] Nuno-Solinis R, Rodriguez-Pereira C, Pinera-Elorriaga K, Zaballa-Gonzalez I, Bikandi-Irazabal J. [Panorama of self-management initiatives in Spain]. Gac Sanit. 2013 Jul-Aug;27(4):332-7. doi: 10.1016/j.gaceta.2013.01.008. Epub 2013 Mar 5. Spanish. PMID 23465729
- [Derived] Ginel-Mendoza L, Hidalgo-Natera A, Reina-Gonzalez R, Poyato-Ramos R, Morales-Naranjo J, Lupianez-Perez I, Baca-Osorio A, Gutierrez-Jansen M, Fernandez-Lara MP, Lozano-Noriega D, Salgado-Carvallo U, Bandera-Garcia C, Navarro-Moya FJ. Efficacy of a joint didactic intervention using the Junta De Andalucia School for Patients method to control prothrombin time in patients taking anticoagulants: protocol for a randomized controlled trial. Trials. 2021 Jan 11;22(1):45. doi: 10.1186/s13063-020-04972-1. PMID 33430922
- See also: Registered follow-up of individualized pharmacological treatment in patients with oral anticoagulation — http://cuidados20.san.gva.es/documents/16605/18107/Seguimiento+de+pacientes+anticoagulados.pdf